CLINICAL TRIAL: NCT00313313
Title: A Multicenter, Randomized, Double-Blind Placebo-Controlled Phase 3 Trial to Evaluate the Efficacy and Safety of Saxagliptin in Combination With Glyburide in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control With Glyburide Alone
Brief Title: A Study of Saxagliptin in Subjects With Type 2 Diabetes Who Have Inadequate Blood Sugar Control With Sulfonylureas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV181-040
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Results first posted 2009-09-25 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — saxagliptin; Glyburide; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Saxagliptin 2.5 mg + Glyburide 7.5 mg (A) (Experimental): Metformin 500-2500 mg (as needed)
  Interventions: Drug: Saxagliptin; Drug: Glyburide; Drug: Metformin
- Saxagliptin 5 mg + Glyburide 7.5 mg (B) (Experimental): Metformin 500-2500 mg (as needed)
  Interventions: Drug: Saxagliptin; Drug: Glyburide; Drug: Metformin
- Placebo + Glyburide 7.5 mg (C) (Placebo Comparator): Metformin 500-2500 mg (as needed)
  Interventions: Drug: Placebo; Drug: Glyburide; Drug: Metformin

INTERVENTIONS:
Drug: Saxagliptin — Tablets, Oral, 2.5 mg, Daily AM, (24 weeks short-term [ST], 12 months long-term [LT])
  Other Names: BMS-477118
  Arms: Saxagliptin 2.5 mg + Glyburide 7.5 mg (A)
Drug: Saxagliptin — Tablets, Oral, 5 mg, Daily AM (24 weeks ST, 12 months LT).
  Other Names: BMS-477118
  Arms: Saxagliptin 5 mg + Glyburide 7.5 mg (B)
Drug: Glyburide — Capsules, Oral, OL, 7.5 mg, Daily, AM (24 weeks ST, 12 months LT)
  Arms: Saxagliptin 2.5 mg + Glyburide 7.5 mg (A); Saxagliptin 5 mg + Glyburide 7.5 mg (B)
Drug: Placebo — Tablets, Oral, 0 mg, Daily AM/PM, (24 weeks ST, 12 months LT)
  Arms: Placebo + Glyburide 7.5 mg (C)
Drug: Glyburide — Capsules, Oral, DB Glyburide, 2.5 mg titrated to 7.5 mg + 7.5 mg OL, Daily AM/PM (24 weeks ST, 12 months LT)
  Arms: Placebo + Glyburide 7.5 mg (C)
Drug: Metformin — Tablets, Oral, OL, 500 - 2500 mg, 1 or 2 times per day (12 months LT)

SUMMARY:
The purpose of this trial is to understand if adding saxagliptin to a sulfonylurea is safe and works better than increasing the amount of sulfonylurea a patient takes

DETAILED DESCRIPTION:
All subjects will participate in a lead-in period, and qualifying subjects will continue into a short-term randomized treatment period. Subjects who complete the short-term period will be eligible to enter the long term extension period. Also, subjects in the short-term period who have an elevated blood sugar that requires additional medication for blood sugar control (defined as rescue) will be eligible to enter the long-term treatment extension period where they will receive metformin.Rescue treatment with metformin is also available during the long-term extension period for subjects who meet glycemic criteria.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes.
* Treated with a sulfonylurea for at least 2 months.
* Inadequate blood sugar control.
* Are not on any other medications to lower blood sugar.
* No major heart, liver or kidney problems.
* Women not pregnant or breast feeding.

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Actual)
Dates: Start 2006-04; Primary Completion 2007-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (103):
- United States (54):
  - Reserach Solutions, Llc, Jonesboro, Arkansas
  - Searcy Medical Center, Searcy, Arkansas
  - Stewart Medical Group, Alhambra, California
  - Southland Clinical Research Center, Inc., Fountain Valley, California
  - Valley Research, Fresno, California
  - Randall Shue, D.O., Los Angeles, California
  - Clinical Trials Research, Roseville, California
  - New West Physicians, Golden, Colorado
  - Phoenix Internal Medicine Associates, Llc, Waterbury, Connecticut
  - Christiana Care Research Institute, Newark, Delaware
  - Central Florida Clinical Trials, Altamonte Springs, Florida
  - Family Care Assoc & Emerald Care Res Grp, Chipley, Florida
  - Clinical Therapeutics Corporation, Coral Gables, Florida
  - Fpa Clinical Research, Kissimmee, Florida
  - Emerald Coast Research Group, Marianna, Florida
  - University Of Miami Diabetes Research Inst., Miami, Florida
  - Atlanta Pharmaceutical Research Center, Inc, Dunwoody, Georgia
  - Cedar-Crosse Research Ctr, Chicago, Illinois
  - Family Medical Center Of Hart Co., Munfordville, Kentucky
  - Columbia Medical Practice, Columbia, Maryland
  - Va Medical Center, Kansas City, Missouri
  - St. Louis Center For Clinical Research, St Louis, Missouri
  - Nevada Alliance Against Diabetes, North Las Vegas, Nevada
  - Physicians Research Center, Toms River, New Jersey
  - Cny Family Care, East Syracuse, New York
  - Metrolina Internal Medicine, Charlotte, North Carolina
  - Med Res Assoc Charlotte, Charlotte, North Carolina
  - Regional Physicians Research, High Point, North Carolina
  - Diabetes & Endocrinology Consultants, Pc, Morehead City, North Carolina
  - Mountain Top Clinical Research Center, Sparta, North Carolina
  - Daystar Clinical Research, Inc., Akron, Ohio
  - Community Health Care, Canal Fulton, Ohio
  - Triphase Research, Ltd., Franklin, Ohio
  - Albert J Weisbrot,Md&Assoc Inc, Mason, Ohio
  - Dr Bahagwan Dass Md, Youngstown, Ohio
  - Oklahoma Cardiovascular And Hypertension Center, Oklahoma City, Oklahoma
  - Utica Park Clinic, Tulsa, Oklahoma
  - Integris Family Care Yukon, Yukon, Oklahoma
  - Coordinators Plus, Llc, Eugene, Oregon
  - Oregon Clinical Research, Portland, Oregon
  - Pearl Clinical Research, Norristown, Pennsylvania
  - Banksville Medical Pc, Pittsburgh, Pennsylvania
  - Guthrie Clinic, Ltd, Sayre, Pennsylvania
  - Upstate Pharmaceutical Research, Simsonville, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Southeastern Research Assoc, Taylors, South Carolina
  - Capital Medical Clinic, Llp, Austin, Texas
  - Texas Center For Drug Development, P.A., Houston, Texas
  - Breath Of Life Research Institute, Katy, Texas
  - Diabetes & Glandular Disease Research Assoc, Pa, San Antonio, Texas
  - S.A.M. Clinical Research Center, San Antonio, Texas
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Office Of Dr. Gray, Spokane, Washington
  - Advanced Healthcare S.C., Milwaukee, Wisconsin
- Argentina (3):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
- Brazil (9):
  - Local Institution, B. Rodolfo Teofilo, Ceará
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Belém, Pará
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Campinas, São Paulo
  - Local Institution, Marília, São Paulo
  - Local Institution, Sao Paulo - Sp, São Paulo
  - Local Institution, Vila Mariana, São Paulo
- Hong Kong (2):
  - Local Institution, Hong Kong
  - Local Institution, Kowloon
- Israel (8):
  - Local Institution, Giv‘atayim
  - Local Institution, Haifa
  - Local Institution, Holon
  - Local Institution, Jerusalem
  - Local Institution, Rishon LeZiyyon
  - Local Institution, Safed
  - Local Institution, Tel Aviv
  - Local Institution, Ẕerifin
- Mexico (7):
  - Local Institution, Durango, Durango
  - Local Institution, Tijuana, B.C., Estado de Baja California
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Df, Mexico City
  - Local Institution, Cuernavaca, Morelos
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Mérida, Yucatán
- Peru (2):
  - Local Institution, Lima, Lima Province
  - Local Institution, San Isidro, Lima region
- Philippines (3):
  - Local Institution, Cebu
  - Local Institution, Manila
  - Local Institution, Quezon
- Puerto Rico (3):
  - Local Institution, Carolina
  - Local Institution, Guaynabo
  - Local Institution, Ponce
- Local Institution, Singapore, Singapore
- South Africa (5):
  - Local Institution, Umhlanga, KwaZulu-Natal
  - Local Institution, Kimberley, Northern Cape
  - Local Institution, Tygerberg, Western Cape
  - Local Institution, Cape Town
  - Local Institution, Johannesburg
- South Korea (3):
  - Local Institution, Kyunggi-Do
  - Local Institution, Seoul
  - Local Institution, Suwon
- Taiwan (3):
  - Local Institution, Changhua
  - Local Institution, Taichung
  - Local Institution, Taipei

REFERENCES:
- [Background] Chacra AR, Tan GH, Apanovitch A, Ravichandran S, List J, Chen R; CV181-040 Investigators. Saxagliptin added to a submaximal dose of sulphonylurea improves glycaemic control compared with uptitration of sulphonylurea in patients with type 2 diabetes: a randomised controlled trial. Int J Clin Pract. 2009 Sep;63(9):1395-406. doi: 10.1111/j.1742-1241.2009.02143.x. Epub 2009 Jul 15. PMID 19614786
- [Derived] Perl S, Cook W, Wei C, Iqbal N, Hirshberg B. Saxagliptin Efficacy and Safety in Patients With Type 2 Diabetes and Moderate Renal Impairment. Diabetes Ther. 2016 Sep;7(3):527-35. doi: 10.1007/s13300-016-0184-9. Epub 2016 Jul 11. PMID 27402391
- [Derived] Bonora E, Bryzinski B, Hirshberg B, Cook W. A post hoc analysis of saxagliptin efficacy and safety in patients with type 2 diabetes stratified by UKPDS 10-year cardiovascular risk score. Nutr Metab Cardiovasc Dis. 2016 May;26(5):374-9. doi: 10.1016/j.numecd.2015.11.004. Epub 2015 Dec 1. PMID 27033025
- [Derived] Karyekar CS, Frederich R, Ravichandran S. Clinically relevant reductions in HbA1c without hypoglycaemia: results across four studies of saxagliptin. Int J Clin Pract. 2013 Aug;67(8):759-67. doi: 10.1111/ijcp.12212. Epub 2013 Jun 24. PMID 23795975
- [Derived] Karyekar C, Donovan M, Allen E, Fleming D, Ravichandran S, Chen R. Efficacy and safety of saxagliptin combination therapy in US patients with type 2 diabetes. Postgrad Med. 2011 Jul;123(4):63-70. doi: 10.3810/pgm.2011.07.2305. PMID 21680990
- [Derived] Chacra AR, Tan GH, Ravichandran S, List J, Chen R; CV181040 Investigators. Safety and efficacy of saxagliptin in combination with submaximal sulphonylurea versus up-titrated sulphonylurea over 76 weeks. Diab Vasc Dis Res. 2011 Apr;8(2):150-9. doi: 10.1177/1479164111404574. PMID 21562067

RESULTS

PARTICIPANT FLOW:
Groups:
- Saxagliptin 2.5 mg + Glyburide 7.5 mg: The Saxagliptin 2.5 mg + Glyburide 7.5 mg group includes data from subjects randomized to receive coadministration of blinded saxagliptin 2.5 mg oral tablets and open-label glyburide 7.5 mg oral tables once daily. Open-label glyburide may have been down titrated by 2.5 mg once due to hypoglycemia as deemed necessary by the investigator.
- Saxagliptin 5 mg + Glyburide 7.5 mg: The Saxagliptin 5 mg + Glyburide 7.5 mg group includes data from subjects randomized to receive coadministration of blinded saxagliptin 5 mg oral tablets and open-label glyburide 7.5 mg oral tables once daily. Open-label glyburide may have been down titrated by 2.5 mg once due to hypoglycemia as deemed necessary by the investigator.
- Placebo + Glyburide 7.5 mg: The Placebo + Glyburide 7.5 mg group includes data from subjects randomized to receive coadministration of blinded placebo oral tablets, blinded glyburide 2.5 mg, and open-label glyburide 7.5 mg once daily. Open-label glyburide may have been down titrated by 2.5 mg once due to hypoglycemia as deemed necessary by the investigator. Blinded glyburide may have been uptitrated by 5 mg according to glycemic criteria provided it had not been previously down-titrated.
Period: Overall Study
Arm/Group | Saxagliptin 2.5 mg + Glyburide 7.5 mg | Saxagliptin 5 mg + Glyburide 7.5 mg | Placebo + Glyburide 7.5 mg
Started | 248 | 253 | 267
Completed | 185 (61 subjects completed the study without being rescued) | 187 (55 subjects completed the study without being rescued) | 185 (26 subjects completed the study without being rescued)
Not Completed | 63 | 66 | 82
Not completed — Lack of Efficacy | 14 | 9 | 20
Not completed — Withdrawal of consent by subject | 18 | 17 | 31
Not completed — Lost to Follow-up | 10 | 7 | 9
Not completed — Adverse Event | 15 | 16 | 12
Not completed — Physician Decision | 2 | 6 | 4
Not completed — Poor/Noncompliance | 3 | 6 | 2
Not completed — Pregnancy | 1 | 2 | 0
Not completed — Death | 0 | 0 | 2
Not completed — Subject No Longer Meets Study Criteria | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin 2.5 mg + Glyburide 7.5 mg | Saxagliptin 5 mg + Glyburide 7.5 mg | Placebo + Glyburide 7.5 mg | Total
Number analyzed (Participants) | 248 | 253 | 267 | 768
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.36 (9.58) | 54.85 (9.96) | 55.06 (10.69) | 55.09 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 143 | 144 | 422
  Male | 113 | 110 | 123 | 346

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (A1C) at Week 24
Description: Mean change from baseline in A1C at Week 24, adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in analysis of change from baseline to Week 24 Last Observation Carried Forward (LOCF), participants must have had a baseline and at least 1 post-baseline measurement. If participant received rescue medication, measurement must have been taken before rescue.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Saxagliptin 2.5 mg + Glyburide 7.5 mg | Saxagliptin 5 mg + Glyburide 7.5 mg | Placebo + Glyburide 7.5 mg
Number analyzed (Participants) | 246 | 250 | 264
percent
  Baseline Mean | 8.36 (0.057) | 8.48 (0.056) | 8.44 (0.055)
  Week 24 Mean | 7.83 (0.074) | 7.83 (0.074) | 8.52 (0.077)
  Adjusted Mean Change from Baseline | -0.54 (0.059) | -0.64 (0.059) | 0.08 (0.057)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Mean change from baseline in FPG at Week 24, adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in analysis of change from baseline to Week 24 LOCF, participants must have had a baseline and at least 1 post-baseline measurement. If a participant received rescue medication, then that measurement must have been taken before rescue.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg + Glyburide 7.5 mg | Saxagliptin 5 mg + Glyburide 7.5 mg | Placebo + Glyburide 7.5 mg
Number analyzed (Participants) | 247 | 252 | 265
mg/dL
  Baseline Mean | 170.1 (2.67) | 175.0 (2.79) | 174.4 (2.64)
  Week 24 Mean | 164.4 (2.76) | 164.6 (2.76) | 174.6 (2.93)
  Adjusted Mean Change from Baseline | -7.1 (2.42) | -9.7 (2.39) | 0.7 (2.33)

3. Secondary Outcome: Percentage of Participants Achieving A1C < 7% at Week 24
Description: Percentage of participants achieving A1C < 7%, the American Diabetes Association's defined goal for glycemia, at each dose of saxagliptin plus glyburide versus placebo plus upward titrated glyburide at Week 24.
Time Frame: Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in the Week 24 LOCF analysis, participants must have had at least 1 post-baseline measurement. If a participant received rescue medication, then that measurement must have been taken before rescue.
Measure: Number; unit: Percentage of participants
Arm/Group | Saxagliptin 2.5 mg + Glyburide 7.5 mg | Saxagliptin 5 mg + Glyburide 7.5 mg | Placebo + Glyburide 7.5 mg
Number analyzed (Participants) | 246 | 250 | 264
Percentage of participants | 22.4 | 22.8 | 9.1

4. Secondary Outcome: Changes From Baseline in Postprandial Glucose (PPG) Area Under the Curve (AUC) Response to an Oral Glucose Tolerance Test (OGTT) at Week 24
Description: Mean change from baseline for 0 to 180 minutes PPG AUC at Week 24, adjusted for baseline values.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg*min/dL
Arm/Group | Saxagliptin 2.5 mg + Glyburide 7.5 mg | Saxagliptin 5 mg + Glyburide 7.5 mg | Placebo + Glyburide 7.5 mg
Number analyzed (Participants) | 190 | 195 | 204
mg*min/dL
  Baseline Mean | 49124 (677.2) | 50342 (669.0) | 51801 (656.9)
  Week 24 Mean | 45402 (681.5) | 45391 (699.3) | 52416 (703.7)
  Adjusted Mean Change from Baseline | -4296 (595.0) | -5000 (585.5) | 1196 (574.5)

ADVERSE EVENTS:
Arm/Group | Placebo + Glyburide 7.5 mg | Saxagliptin 2.5 mg + Glyburide 7.5 mg | Saxagliptin 5 mg + Glyburide 7.5 mg
Serious Adverse Events (participants affected / at risk) | 23/267 | 18/248 | 12/253
Other Adverse Events (participants affected / at risk) | 163/267 | 144/248 | 154/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Glyburide 7.5 mg (N=267) | Saxagliptin 2.5 mg + Glyburide 7.5 mg (N=248) | Saxagliptin 5 mg + Glyburide 7.5 mg (N=253)
ANGINA PECTORIS (Cardiac disorders) | 1 | 0 | 0
CARDIOGENIC SHOCK (Cardiac disorders) | 0 | 0 | 1
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 2 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 1 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 | 0 | 1
EXTREMITY NECROSIS (Vascular disorders) | 0 | 0 | 1
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 2
SYNCOPE (Nervous system disorders) | 1 | 0 | 0
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 1 | 0
ASCITES (Gastrointestinal disorders) | 0 | 1 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 0
SALIVARY GLAND MASS (Gastrointestinal disorders) | 0 | 0 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 1 | 1
PNEUMONIA (Infections and infestations) | 3 | 0 | 0
APPENDICITIS (Infections and infestations) | 0 | 2 | 0
PYELONEPHRITIS (Infections and infestations) | 1 | 0 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 1 | 0
WOUND INFECTION (Infections and infestations) | 1 | 0 | 0
CELLULITIS ORBITAL (Infections and infestations) | 0 | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 3 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 1
GASTROINTESTINAL INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
ASTHENIA (General disorders) | 0 | 1 | 0
CHEST PAIN (General disorders) | 0 | 2 | 0
SUDDEN CARDIAC DEATH (General disorders) | 1 | 0 | 0
ADENOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Glyburide 7.5 mg (N=267) | Saxagliptin 2.5 mg + Glyburide 7.5 mg (N=248) | Saxagliptin 5 mg + Glyburide 7.5 mg (N=253)
HYPERTENSION (Vascular disorders) | 15 | 15 | 23
HEADACHE (Nervous system disorders) | 23 | 23 | 25
DIARRHOEA (Gastrointestinal disorders) | 27 | 22 | 16
DYSPEPSIA (Gastrointestinal disorders) | 8 | 13 | 10
GASTRITIS (Gastrointestinal disorders) | 9 | 13 | 8
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 | 16 | 7
INFLUENZA (Infections and infestations) | 27 | 21 | 19
PHARYNGITIS (Infections and infestations) | 15 | 11 | 19
NASOPHARYNGITIS (Infections and infestations) | 29 | 21 | 26
PHARYNGOTONSILLITIS (Infections and infestations) | 11 | 13 | 5
URINARY TRACT INFECTION (Infections and infestations) | 32 | 33 | 42
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 25 | 17 | 24
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 12 | 11 | 13
BACK PAIN (Musculoskeletal and connective tissue disorders) | 18 | 18 | 16
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 20 | 18 | 20
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 19 | 14 | 15
COUGH (Respiratory, thoracic and mediastinal disorders) | 17 | 19 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.